CLINICAL TRIAL: NCT06863766
Title: Effects of Daily Supplementation With Milk Powder on Blood Glucose Control and Fluctuation in Middle-aged and Older Adults: A Randomized Control Trial
Brief Title: Effects of Milk Powder Intervention on Blood Glucose Control and Fluctuation in Middle-aged and Elderly People With Pre-diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huilian Zhu (Other)
Responsible Party: Sponsor-Investigator, Huilian Zhu, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MN-2024-07
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- fortified formula milk powder group (Experimental): Fortified formula milk powder is supplemented with fiber, bitter gourd powder,mulberry leaves extract, whitekidney beans extract, and probiotics, and packaged in 25-gram sachets. The milk powder is consumed orally, two sachets per day for a duration of 8 weeks.
  Interventions: Dietary Supplement: fortified formula milk powder group
- regular milk powder group (Placebo Comparator): Regular milk powder does not contain and additional supplementation, and the color, flavor, shape, taste, and weight are same with the formula milk powder.
  Interventions: Dietary Supplement: regular milk powder group

INTERVENTIONS:
Dietary Supplement: fortified formula milk powder group — Fortified formula milk powder is supplemented with fiber, bitter gourd powder,mulberry leaves extract, whitekidney beans extract, and probiotics, and packaged in 25-gram sachets. The milk powder is consumed orally, two sachets per day for a duration of 8 weeks.
  Arms: fortified formula milk powder group
Dietary Supplement: regular milk powder group — Regular milk powder does not contain and additional supplementation, and the color, flavor, shape, taste, and weight are same with the formula milk powder.
  Arms: regular milk powder group

SUMMARY:
This study aims to conduct a 8-week intervention involving one formula milk powder for middle-aged and elderly individuals with pre-diabetes, assessing its impact on blood glucose control and fluctuations in comparison to interventions using regular milk powder.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 75 years, regardless of gender.
2. Impaired fasting glucose (5.6 mmol/L ≤ FPG < 6.9 mmol/L) or glycated hemoglobin (HbA1c) between 5.7-6.4% (39-47 mmol/mol).
3. Resided in Guangzhou for the past six months and no plans to relocate or travel outside the city in the next month.
4. Signed informed consent form and voluntarily agreed to participate in the project.

Exclusion Criteria:

1. Patients with a confirmed diagnosis of diabetes who are currently taking glucose-lowering medications (e.g., insulin, GLP-1 receptor agonists, or SGLT2 inhibitors).
2. Individuals with lactose intolerance or dairy product intolerance.
3. Pregnant, planning to become pregnant within the next three months, or currently breastfeeding.
4. Weight change > 5% in the past three months or plans to lose weight or change dietary habits.
5. Alcohol consumption > 40g/day.
6. Individuals with communication barriers, cognitive impairments, or other conditions that may prevent them from completing the study procedures.
7. Severe diseases that may affect participation in the study, including but not limited to endocrine disorders, severe cardiovascular or cerebrovascular diseases, cancer, metabolic diseases, etc.
8. Participation in or current involvement in other clinical trials within the past three months.
9. No use of antibiotic medications within the past three months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
fasting blood glucose | up to 8 weeks
  At baseline, and 8 weeks, investigators will use automatic electrochemiluminescence analyzer to examine fasting blood glucose.
2h-piAUC after standardized breakfast | up to 8 weeks
  the positive increment of area under curve in 2 hours after standardized breakfast standardized breakfast, measured by continuous glucose monitoring at baseline, and 8 weeks.
TIR (time in range) | up to 8 weeks
  TIR refers to the time when blood glucose is controlled within a reasonable ( target ) range (3.9~10.0 mmol/L), measured by continuous glucose monitoring at baseline and 8 weeks.

SECONDARY OUTCOMES:
HbA1c | up to 8 weeks
  At baseline, and 8 weeks, investigators will use automatic electrochemiluminescence analyzer to examine HbA1c.
weight | up to 8 weeks
  At baseline, and 8 weeks, investigators will examine weight.
intestinal bacteria | up to 8 weeks
  At baseline, and 8 weeks, investigators will use 16S rRNA pyrosequencing to examine intestinal bacteria.
lipid metabolism | up to 8 weeks
  At baseline, and 8 weeks, investigators will use automatic electrochemiluminescence analyzer to examine total cholesterol, low density lipoprotein, high density lipoprotein, triglyceride.
sleep quality | up to 8 weeks
  At baseline, and 8 weeks, investigators will use the Pittsburgh sleep quality index scale to examine sleep quality.
blood pressure | up to 8 weeks
  At baseline, and 8 weeks, investigators will test the systolic blood pressure and diastolic blood pressure using automatic digital blood pressure monitor
Continuous Glucose Monitoring (CGM) Data | up to 8 weeks
  At baseline, and 8 weeks, investigators will using Continuous Glucose Monitoring (CGM) to monitor the glucose level of participants

IPD SHARING:
Plan to Share IPD: No